CLINICAL TRIAL: NCT03419572
Title: Prospective Non Interventional Study of Cabozantinib Tablets in Adults With Advanced Renal Cell Carcinoma Following Prior Vascular Endothelial Growth Factor (VEGF)-Targeted Therapy
Brief Title: Non-interventional Study of Cabozantinib in Adults With Advanced Renal Cell Carcinoma
Acronym: CASSIOPE
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: F-FR-60000-001; EUPAS19464 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2017-12-15; First posted 2018-02-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Second line therapy: Data collection
  Interventions: Other: Data collection
- Third and later line therapy: Data collection
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Only available evaluations as decided by the investigator based on local clinical practice will be collected.

SUMMARY:
The objective of this study is to understand the utilization of cabozantinib in subjects with advanced renal cell carcinoma (RCC) following prior VEGF-targeted therapy in real life settings in terms of dose modifications due to adverse events (AEs) when used as a second line therapy or third and later line therapy. Other patterns of use of cabozantinib will also be described.

DETAILED DESCRIPTION:
The study will follow the real-life management of patients in clinical practice. Visits will take place according to the study site's clinical practice. Cabozantinib is to be administered as directed by the investigator according to the study site's usual clinical practice and the Cabometyx™ Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Has a diagnosis of advanced RCC
* Has received at least one prior VEGF-targeted therapy
* For whom the treating physician has decided to start treatment with cabozantinib tablets prior to inclusion
* No previous exposure to cabozantinib prior to inclusion
* Not concurrently involved in an interventional study
* Consents to participate in this noninterventional study

Exclusion Criteria:

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with advanced RCC following prior VEGF-targeted therapy in real life settings.
Sampling Method: Non-Probability Sample
Enrollment: 689 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with dose modifications due to AEs | 12 months

SECONDARY OUTCOMES:
Reason for cabozantinib dose modification (any modification, reduction, temporary interruption or discontinuation) | 12 months
  Percentage of subjects with the following reasons - Disease progression, Adverse event, Subject non-compliance, Treatment resumed or re escalated, Subject decision, Clinical / investigator decision, Other
Description of number of cabozantinib dose modifications (any modification, reduction, temporary interruption, increase or discontinuation) | 12 months
Median time to first cabozantinib dose modification (any modification, reduction, temporary interruption, increase or discontinuation) due to AEs and for any reason | 12 months
Description of cabozantinib starting dose (combination of dose per intake and frequency) | 12 months
Description of daily dose of cabozantinib received | 12 months
Description of cabozantinib dose intensity (average daily dose compared to starting dose) | 12 months
Duration of cabozantinib treatment (expressed as mean and median time to end of treatment) | 12 months
Proportion of subjects with concomitant radiotherapies | 12 months
Description of systemic therapy (drug name) planned following cabozantinib discontinuation | 12 months
  Percentage of subjects treated with the following drugs: Sunitinib, Pazopanib, Axitinib, Sorafenib, Bevacizumab, Cytokines, Everolimus, Lenvatinib, Nivolumab, Tivozanib, Experimental trial drug, Other, Unknown)
Overall best response | 12 months
  Per investigator assessment
Median Progression Free Survival (PFS) time | 12 months
  Defined as the time between the start date of cabozantinib and the date of progression or death. Clinical and radiographic (assessed by the investigator based on RECIST 1.1)
Overall Survival (OS) rate at the end of the study | 12 months
Health care resource utilisation: number of visits to health care professionals (hospitalisation, surgical procedure, emergency room, physician, homecare by nurse) associated with the management of treatment-related AEs | 12 months
Health care resource utilisation: Description of concomitant medications (by drug class and preferred name) associated with the management of treatment-related AEs | 12 months
Health care resource utilisation: Description of number of unplanned laboratory tests associated with the management of treatment-related AEs | 12 months

OTHER OUTCOMES:
Incidence of all treatment-emergent non-serious and serious AEs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (91):
- Austria (2):
  - Kepler University Hospital - Urology, Linz
  - Universitatsklinikum fur Urologie und Andrologie, Salzburg
- Belgium (5):
  - Imelda Ziekenhuis, Bonheiden
  - Az Klina, Brasschaat
  - UZA, Edegem
  - Jessa Ziekenhuis, Hasselt
  - Az Damiaan, Ostend
- Czechia (4):
  - Krajská Nemocnice Liberec, A.S., Komplexní Onkologické Centrum, Liberec
  - Fakultni Nemocnice Kralovske Vinohrady (FNKV) - Radioterapeuticka a Onkologicka klinika, Prague
  - Thomayerova Nemocnice, Onkologická Klinika 1. LF UK A TN, Prague
  - Fakultni Nemocnice na Bulovce, Institut of Radiation Oncology, Prague
- France (16):
  - CHU Angers, Angers
  - CH Cote Basque, Bayonne
  - Centre Hospitalier Universitaire, Besançon
  - Hopital Saint Andre - CHU de Bordeaux, Bordeaux
  - Centre Catalan d'Urologie, Cabestany
  - Centre Maurice Tubiana, Caen
  - CHU Henri Mondor, Créteil
  - Grenoble University Hospital, Grenoble
  - Polyclinique Chénieux, Limoges
  - L'institut Mutualiste Montsouris, Paris
  - Hospital De Cornouaille, Quimper
  - Centre de Lutte Contre le Cancer (CLCC) - Institut Jean Godinot, Reims
  - Institut de Cancérologie Lucien Neuwirth (ICLN), Saint-Priest-en-Jarez
  - Strasbourg Oncologie Liberale, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Tours - Hopital Bretonneau, Tours
- Germany (11):
  - Vivantes Klinikum Neukolln, Berlin
  - MVZ- Polyclinic Eisenach, Eisenach
  - Universitaetsklinikum Frankfurt - Department of Urology, Frankfurt
  - University Medical Center Halle (Saale), Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Asklepios Clinic Altona Hamburg, Hamburg
  - University Medical Center LMU Munich - Campus Grosshadern, Urologische Klinik und Poliklinik Marchionnish R. 15, München
  - Universitätsklinikum Münster, Münster
  - MVP MP Saaletal Saalfeld/Saale, Saalfeld
  - Dept of Urology, Eberhard-Karls-University Tuebingen, Tübingen
  - University Medical Center Ulm, Ulm
- Greece (7):
  - Evaggelismos Hospital, Athens
  - Saint Savvas Hospital, Athens
  - Alexandra Hospital, Athens
  - G.O.H.K "Oi Agioi Anargiroi", Athens
  - Dep. Medical Oncology, University Hospital of Ioannina, Ioannina
  - Papageorgiou Hospital, Thessaloniki
  - Interbalkan Medical Center, Thessaloniki
- Italy (14):
  - Azienda Ospedaliera S.Orsola Malpighi di Bologna, Bologna
  - Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Aorn Cardarelli, Napoli
  - National Cancer Institute "Fondazione G. Pascale" IRCCS, Napoli
  - Umberto Basso, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Fondazione Salvatore Maugeri - I.R.C.C.S, Pavia
  - IRCCS Azienda Usl Di Reggio Emilia, Reggio Emilia
  - Gemelli Hospital, Roma
  - UOC Oncologia Azienda Ospedaliera Sant-Andrea, Rome
  - Presidio Ospedaliero Santa Chiara, Trento
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
  - San Bortolo General Hospital, Vicenza
- Netherlands (4):
  - Amphia Ziekenhuis, Breda
  - Deventer Hospital, Deventer
  - Haaglanden Medical Centre, Leidschendam
  - Franciscus Gasthuis Hospital, Rotterdam
- Poland (5):
  - Onkology Center, Bydgoszcz
  - Szpital Kliniczny Przemienienia Panskiego w Poznaniu, Poznan
  - Magodent SP Z O.O., Warsaw
  - Wojskowy Instytut Medyczny, Klinika Onkologii, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Spain (17):
  - Hospital Vall de Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Dr. Josep Trueta, Girona
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Ramón y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias (Huca), Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Complejo Hospitalario De Navarra, Pamplona
  - Hospital Universitari Parc Tauli, Sabadell
  - Complejo Hospitalario Universitario de Compostela, Santiago de Compostela
  - Hospital Álvaro Cunqueiro de Vigo, Vigo
  - Hospital Clinico Lozano Blesa de Zaragoza, Zaragoza
- United Kingdom (6):
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Royal Derby Hospital, Derby
  - Freeman Hospital-Northern Centre For Cancer Care, Newcastle
  - Mount Vernon Cancer Centre - East and North Hertfordshire NHS Trust, Northwood
  - Rosemere Cancer Centre, Royal Preston Hospital, Preston
  - Frimley Health NHS Foundation Trust - Wezham Park and Heatherwood Hospitals, Slough